CLINICAL TRIAL: NCT01421940
Title: The Efficacy of Penile Rehabilitation Using Udenafil After Total Mesorectal Excision of Rectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Colorectal Cancer Center, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KNUHCRC002
Record Dates: First submitted 2011-08-01; First posted 2011-08-23 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Rectal Cancer
Keywords: Udenafil; rectal cancer; penile rehabilitation; total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Individuals who take placebo after total mesorectal excision
  Interventions: Drug: Placebo drug
- Udenafil (Experimental): Individuals who take udenafil after total mesorectal excision
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Placebo drug — After total mesorectal excision for rectal cancer, patients take placebo drug five time per week for 12 weeks.
  Arms: Control
Drug: Udenafil — After total mesorectal excision, patients take 50mg udenafil five times per week for 12 weeks.
  Arms: Udenafil

SUMMARY:
Sexual dysfunctions are well-recognized complications after rectal cancer surgery. Damage to the pelvic plexus and pelvic splanchnic nerves results in ejaculatory dysfunction. The purpose of this study is to evaluate the efficacy of Udenafil(Zydena®, Dong-A Pharmaceutical co., Ltd, Seoul, Korea) in penile rehabilitation for patients who undertake total mesorectal excision.

ELIGIBILITY:
Inclusion Criteria:

* Age : 20-65
* Rectal cancer within 15cm from anal verge
* Patients with more than 5 points decreased IIEF-5 after operation
* Patients with sexual activity

Exclusion Criteria:

* Preoperative IIEF-5 : ≤14
* Recent MI, CVA, nitrate medication
* Severe cardiovascular disease, psychiatric disease
* Severe hepatic dysfunction (GOT, GPT ≥100IU/L)
* Renal dysfunction (Cr ≥2mg/dl)

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in International Index of Erectile Function (5-item Version) at 12 and 24 week | Baseline, 12weeks, 24 weeks
  * IIEF-5 questionnaire is used to assess male erectile function
  * IIEF-5 (5-item Version of the International Index of Erectile Function)is obtained by combining the scores of the responses to 5 questions. Each question is scored from 0-5 (1 questions is scored from 1-5) for IIEF-5 range of 1-25 points; lower numerical scores from the IIEF-5 questionnaire represnt greater severitt of erectile dysfunction.

SECONDARY OUTCOMES:
Change from baseline in SEP Q2,Q3 and GEQ | baseline, 12weeks, and 24 weeks
  * SEP Q2 (Sexual encounter profile Q2) and SEP Q3 (Sexual encounter profile Q3) are used to assess erectile function
  * The efficaty of medication is followed by GEQ (Global efficacy question).
Number of patients with adverse events during 24 weeks of the study | Baseline through 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Medical Center, Daegu, South Korea

REFERENCES:
- [Derived] Park SY, Choi GS, Park JS, Kim HJ, Park JA, Choi JI. Efficacy and safety of udenafil for the treatment of erectile dysfunction after total mesorectal excision of rectal cancer: a randomized, double-blind, placebo-controlled trial. Surgery. 2015 Jan;157(1):64-71. doi: 10.1016/j.surg.2014.07.007. PMID 25482466